CLINICAL TRIAL: NCT01443416
Title: An Alternative Booster Vaccine Against Meningitis and Ear Infections.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVG 2011/05
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Invasive Streptococcus Pneumoniae Disease
Keywords: pneumococcal conjugate vaccine; invasive pneumococcal disease; vaccination; children
MeSH Terms: interventions — 10-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 13-valent pneumococcal conjugate vaccine (Experimental): 12 month booster dose of Prevenar
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- 10-valent pneumococcal conjugate vaccine (Experimental): 12 month booster dose of Synflorix
  Interventions: Biological: 10-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — The vaccine will be given to 12 month old children who have had 2 doses of Prevenar at 2 and 4 months of age
  Arms: 13-valent pneumococcal conjugate vaccine
Biological: 10-valent pneumococcal conjugate vaccine — The vaccine will be given to 12 month old children who have had 2 doses of Prevenar at 2 and 4 months of age.
  Arms: 10-valent pneumococcal conjugate vaccine

SUMMARY:
This is a study to evaluate an alternative booster for pneumococcal conjugate vaccination (PCV) for children at 12 months of age. Currently in the UK, 3 doses of a vaccine called Prevenar 13 (PCV-13), which contains 13 pneumococcal serotypes attached to a carrier protein called CRM197, are given to children at 2, 4 and 12 months of age. There is some evidence that a vaccine called Synflorix (PHiD-CV) may be at least as good as the currently used vaccine when used as an alternative vaccine at 12 months of age. Although PHiD-CV contains only 10 serotypes, there is evidence that it generates cross-reactive antibodies against two of the three additional serotypes included in PCV-13 which might be enough to protect children against disease caused by these two serotypes. Furthermore, previous studies have shown that PHiD-CV confers protection against a common otitis media pathogen in children called nontypeable H. influenzae (NTHi) by attachment to a carrier protein called Protein D, which is derived from NTHi. In addition, the use of a carrier protein, which is not closely related to an antigen included in any coadministered or previously administered routine vaccine minimises the risk of interference related to it.

The investigators aim to recruit 168 healthy children at the age of 12 months who have already received two doses of PCV-13 according to the UK routine immunisation schedule at 2 and 4 months of age. Participants will then be randomised to receive a booster dose of either PCV-13 or PHiD-CV at 12 months of age.

Three visits will take place at their parents' home and will involve a blood test followed by a dose of PCV-13 or PHiD-CV on visit 1, and a blood test on each of the visits 2 (1 month after visit 1) and 3 (1 year after visit 1).

DETAILED DESCRIPTION:
Currently in the UK, 3 doses of a vaccine called Prevenar 13 (PCV-13), which contains 13 pneumococcal serotypes attached to a carrier protein called CRM197, are given to children at 2, 4 and 12 months of age. There is some evidence that a vaccine called Synflorix (PHiD-CV) may be at least as good as the currently used vaccine when used as an alternative vaccine at 12 months of age. Although PHiD-CV contains only 10 serotypes, there is evidence that it generates cross-reactive antibodies against two of the three additional serotypes included in PCV-13 which might be enough to protect children against disease caused by these two serotypes. Furthermore, previous studies have shown that PHiD-CV confers protection against a common otitis media pathogen in children called nontypeable H. influenzae (NTHi) by attachment to a carrier protein called Protein D, which is derived from NTHi. In addition, the use of a carrier protein, which is not closely related to an antigen included in any coadministered or previously administered routine vaccine minimises the risk of interference related to it.

The investigators aim to recruit 168 healthy children at the age of 12 months who have already received two doses of PCV-13 according to the UK routine immunisation schedule at 2 and 4 months of age. Participants will then be randomised to receive a booster dose of either PCV-13 or PHiD-CV at 12 months of age.

Three visits will take place at their parents' home and will involve a blood test followed by a dose of PCV-13 or PHiD-CV on visit 1, and a blood test on each of the visits 2 (1 month after visit 1) and 3 (1 year after visit 1).

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 months (-2 weeks to +6 weeks) at time of enrolment.
* Have received two doses of PCV-13 at less than 6 months of age with a gap of at least 6 weeks between the two vaccinations.
* Have received all primary vaccines according to the UK routine immunisation schedule (up to, but not including, 12 months of age).
* Available for the entire study period and whose parent/legal guardian can be reached by telephone.
* Healthy children as determined by medical history and physical examination, done by a study nurse (and/or study doctor if required, depending on the medical history of the participant and physical assessment), and judgment of the investigator.
* Parent/legal guardian must be able to complete all relevant study procedures during study participation.

Exclusion Criteria:

* Previous receipt of pneumococcal vaccine other than the 13-valent pneumococcal conjugate vaccine (Prevenar 13®, Pfizer).
* Receipt of the routine 12 month immunisations (PCV13 (3rd dose), combined Haemophilus influenzae type b and serogroup C meningococcal glyco-conjugate vaccine (Hib-MenC) or measles, mumps and rubella vaccine (MMR)).
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with pneumococcal conjugate vaccine.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* Known or suspected immune deficiency or suppression.
* History of culture-proven invasive disease caused by S. pneumoniae.
* Major known congenital malformation or serious chronic disorder.
* Significant neurologic disorder or history of seizures including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorder.
* Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies; e.g., Synagis B).
* Parents who plan to move out of the geographical area where the study would be conducted.

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportions of participants who have IgG concentrations ≥0.35mcg/ml for 14 pneumococcal serotypes following vaccination with either Prevenar or Synflorix | One month after a 12 month booster vaccination
  To demonstrate non-inferiority (10% level) of a booster dose of PCV-10 compared to a booster dose of PCV-13 for proportion of participants who have serotype-specific IgG concentrations ≥0.35mcg/ml for the PHiD-CV serotypes (1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, 23F) 1 month following booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, Principal Investigator — University of Oxford
Locations (1):
- Oxford Vaccine Group, Oxford, United Kingdom

REFERENCES:
- [Derived] Truck J, Kelly S, Jawad S, Snape MD, Voysey M, Pollard AJ. Differences in Immunization Site Pain in Toddlers Vaccinated With Either the 10- or the 13-Valent Pneumococcal Conjugate Vaccine. Pediatr Infect Dis J. 2018 Apr;37(4):e103-e106. doi: 10.1097/INF.0000000000001894. PMID 29329169